CLINICAL TRIAL: NCT01463007
Title: ACCELERATED PARTIAL BREAST IRRADIATION USING NON-INVASIVE IMAGE-GUIDED BREAST BRACHYTHERAPY (ACCUBOOST) FOR EARLY STAGE BREAST CANCERS: A TOXICITY ASSESSMENT
Brief Title: Partial Breast Irradiation Using Non Invasive Approach for Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaroslaw Hepel (Other)
Collaborators: The Miriam Hospital (Other); Rhode Island Hospital (Other)
Responsible Party: Sponsor-Investigator, Jaroslaw Hepel, principal investigator, Brown University
Organization: Brown University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 251
Record Dates: First submitted 2011-07-21; First posted 2011-11-01 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: invasive ductal cancer; tubular breast cancer; breast cancer; colloid; ER positive; radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation (Experimental): AccuBoost APBI- 34.0 Gy in 10fx
  Interventions: Radiation: Accelerated partial breast irradiation
- Extended Follow up (Experimental): This arm extends follow up at the Rhode Island Hospital location to 5 years. Annual mammograms and additional documentation is required to be submitted only if completed.
  Interventions: Other: Extended Follow up

INTERVENTIONS:
Radiation: Accelerated partial breast irradiation — Accuboost APBI 34.0 Gy in 10 fractions
  Arms: Radiation
Other: Extended Follow up — This arm extends follow up at the Rhode Island Hospital location to 5 years. Annual mammograms and additional documentation is required to be submitted only if completed.
  Arms: Extended Follow up

SUMMARY:
The purpose of this study is to evaluate the rate of early and intermediate toxicity related to the AccuBoost System for delivery of APBI in women with resected, early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed histological diagnosis of invasive breast carcinoma or DCIS
2. Age greater or equal to 50 years old
3. Life expectancy > 6 months
4. Treated by breast conserving surgery with axillary node dissection or sentinel lymph node biopsy
5. Pathologic tumor size less than or equal to 2 cm
6. Invasive ductal, mucinous, tubular or colloid histology
7. Estrogen receptor positive for invasive carcinoma.
8. Unifocal/unicentric disease
9. Negative surgical margins greater than or equal to 2 mm
10. Pathologic lymph node negative
11. No evidence of lymphovascular invasion
12. ECOG performance status of 0 or 1 (Appendix 1)
13. Informed consent signed.

Exclusion Criteria:

1. Known BRCA 1/2 Mutation; (BRCA 1 and 2 testing is not required)
2. Autoimmune disorder
3. Pregnancy
4. Breast implants
5. Psychiatric or addictive disorder that would preclude attending follow-up
6. Neoadjuvant chemotherapy (adjuvant chemotherapy is permitted)
7. Suspicious remaining microcalcification on post-surgery mammogram (unless biopsy proven benign)
8. Lobular features on histology (pure or mixed) or sarcoma histology
9. Node positive on axillary dissection or in the sentinel lymph node biopsy;
10. Extensive in situ carcinoma (EIC)
11. Multicentric or multifocal disease
12. Paget's disease of the nipple
13. Distant metastases
14. Lumpectomy cavity not well visualized on AccuBoost imaging
15. Lumpectomy cavity with 1cm margin (PTV) not adequately encompassed by any applicator (PTV > 6cm)
16. Breast separation with compression > 7cm.
17. Overlap of skin between orthogonal treatment axes.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09-12 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Hepel, MD, Principal Investigator — Brown University
Locations (4):
- United States (4):
  - Center For Cancer Care and Research- Watson Clinic, Lakeland, Florida
  - Brown University Oncology Research Group, Providence, Rhode Island
  - Lifespan Hospitals, Providence, Rhode Island
  - Tacoma Radiation, Tacoma, Washington

REFERENCES:
- [Derived] Hepel JT, Leonard KL, Sha S, Graves TA, Wiggins DL, Mastras D, Pittier A; Brown University Oncology Research Group; Wazer DE. Phase 2 Trial of Accelerated Partial Breast Irradiation (APBI) Using Noninvasive Image Guided Breast Brachytherapy (NIBB). Int J Radiat Oncol Biol Phys. 2020 Dec 1;108(5):1143-1149. doi: 10.1016/j.ijrobp.2020.07.2312. Epub 2020 Jul 25. PMID 32721422
- [Derived] Hepel JT, Hiatt JR, Sha S, Leonard KL, Graves TA, Wiggins DL, Mastras D, Pittier A; Brown University Oncology Research Group; Wazer DE. The rationale, technique, and feasibility of partial breast irradiation using noninvasive image-guided breast brachytherapy. Brachytherapy. 2014 Sep-Oct;13(5):493-501. doi: 10.1016/j.brachy.2014.05.014. Epub 2014 Jul 3. PMID 24997723

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 patients must COMPLETE treatment. 41 were registered because 1 was removed secondary to Physician decision to not continue treatment.
Period: Overall Study
Arm/Group | Radiation
Started | 41
Completed | 40
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 25
Age, Continuous [Mean (Full Range); unit: years] | 61.46 [50 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Early and Intermediate Toxicity
Description: Any toxicity related to the radiation treatment will be scored and graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 (Appendix 4). Acute side effects are any side effects occurring within 3 months of treatment. Intermediate side effects are any side effects occurring between 3 months and 2 years. This is reported in the outcome table.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Extended to 5 Years of Follow Up-Rhode Island Hospital Only: Follow up has been extended to include follow up visits at 2,6 weeks and at 4,6,12,18,24 months then annually (+/- 6 months) for an additional 3 years for a total of approximately 5 years of follow up.
Arm/Group | Radiation | Extended to 5 Years of Follow Up-Rhode Island Hospital Only
Number analyzed (Participants) | 41 | 28
participants | 40 | 28

2. Secondary Outcome: Cosmetic Outcome
Description: Cosmetic results will be evaluated at each follow-up visit by the treating radiation oncologist using the Harvard criteria inclusive of discomfort during treatment(Pain), Fatigue and Acute skin reaction. This is reported in the outcome table.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Radiation
Number analyzed (Participants) | 41
participants | 35

ADVERSE EVENTS:
Time Frame: Data was collected from signing of ICF until 2 years post treatment.
Arm/Group | Radiation
Serious Adverse Events (participants affected / at risk) | 1/41
Other Adverse Events (participants affected / at risk) | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation (N=41)
Infection (Investigations) | 1 (1)
Creatinine (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Bicarbonate (Investigations) | 1 (1)
SGOT (Investigations) | 1 (1)
Alkaline Phosphatase value (Investigations) | 1 (1)
Hyperbilirubineamia (Investigations) | 1 (1)
Hypoalbuminemia (Investigations) | 1 (1)
Leukocytes (Investigations) | 1 (1)
Hemoglobin (Investigations) | 1 (1)
Neutrophils (Investigations) | 1 (1)
INR (Investigations) | 1 (1)
PTT (Investigations) | 1 (1)
Fibrinogen (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation (N=41)
Discomfort (Investigations) | 35 (35)
acute skin rxn (Investigations) | 32 (32)
skin induration/fibrosis (Investigations) | 11 (11)
hyperpigmentation (Investigations) | 22 (22)
fatigue (Investigations) | 18 (18)
breast volume (Investigations) | 11 (11)
seroma (Investigations) | 2 (2)
fat necrosis (Investigations) | 2 (2)
Itching (Investigations) | 0 (0)
Fibrosis Cosmesis (Investigations) | 1 (1)
Talangiectasis (Investigations) | 8 (8)
breast pain (Investigations) | 7 (7)
Nausea (Investigations) | 1 (1)
Diarrhea (Investigations) | 1 (1)
erythema (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No